CLINICAL TRIAL: NCT06840665
Title: A Prospective, Randomized, Phase II Trial of MR-guided Adaptive Radiotherapy Combined With PD-1 Antibody and CAPOX for Locally Advanced Rectal Cancer
Brief Title: MR-guided Adaptive Radiotherapy Combined With PD-1 Antibody and CAPOX for Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Study Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2024-293-3847
Record Dates: First submitted 2025-02-15; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Locally Advanced Rectal Cancer
MeSH Terms: interventions — spartalizumab; toripalimab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The patients will receive conventional pelvic radiotherapy (30Gy/6Fx), combined with 6 cycles of CAPOX and PD-1 antibody. TME surgery is scheduled after TNT.
  Interventions: Drug: PD-1 antibody; Drug: Oxaliplatin; Drug: Capecitabine
- Group B (Experimental): The patients will receive lymph node-sparing radiotherapy (30Gy/6Fx), combined with 6 cycles of CAPOX and PD-1 antibody. TME surgery is scheduled after TNT.
  Interventions: Drug: PD-1 antibody; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: PD-1 antibody — PD-1 antibody (Toripalimab): 240mg d1 q3w
  Other Names: Toripalimab
Drug: Oxaliplatin — Oxaliplatin: 130mg/m2 d1 q3w
Drug: Capecitabine — Capecitabine: 1000mg/m2 bid d1-14 q3w

SUMMARY:
NeoPulsar is a prospective, randomized phase II trial. 46 LARC (T3-4/N+M0, distance from anal verge ≤12cm) patients will be treated with MR-guided adaptive radiotherapy (30Gy/6Fx) combined with 6 cycles of Toripalimab and CAPOX. TME surgery is scheduled after TNT. The primary endpoint is pathological complete response (pCR) rate. The secondary endpoints include the grade 3-4 acute adverse effects (AE) rate, anal function, surgical complication, 3-year LRFS rate, 3-year DFS rate, 3-year OS rate, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, male or female
2. Pathologically confirmed rectal adenocarcinoma
3. The distance from anal verge ≤ 10 cm
4. Clinical stage T3-4 and/or N+
5. No evidence of distance metastases
6. MSI/MMR status: MSS/pMMR
7. Karnofsky score >=70
8. Adequate organ function and have no contraindications to surgery, radiochemotherapy, or immunotherapy
9. No chemotherapy or any other anti-tumor therapy prior to enrollment
10. No immunotherapy prior to enrollment
11. With good compliance during the study
12. Signed written informed consent

Exclusion Criteria:

1. Known history of other malignancies within 5 years， except cured skin cancer and cervical cancer in situ
2. Pregnancy or breast-feeding women
3. Individuals with a history of uncontrolled epilepsy, central nervous system disease, or psychiatric disorders that, in the judgment of the investigator, are of such clinical severity that they may prevent the signing of an informed consent form or affect the patient's adherence to oral medications
4. Individuals with clinically serious (i.e., active) heart disease, such as symptomatic coronary artery disease, New York Heart Association (NYHA) class II or worse congestive heart failure or severe arrhythmia requiring pharmacologic intervention, or history of myocardial infarction within the last 12 months
5. Individuals with a history of organ transplantation requiring immunosuppressive therapy and long-term hormone therapy
6. Individuals with autoimmune diseases
7. Individuals with severe uncontrolled recurrent infections，or other severe uncontrolled concomitant diseases
8. Baseline hematology and biochemistry not meeting the following criteria: Hb≥90g/L; NEU ≥1.5×109/L; PLT ≥100×109/L; ALT, AST ≤2.5 times the upper limit of normal; ALP ≤2.5 times the upper limit of normal; TB <1.5 times the upper limit of normal; Cr <1 time the upper limit of normal; Alb ≥30g/L
9. Individuals with dihydropyrimidine dehydrogenase (DPD) deficiency
10. Individuals allergic to any drug component of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2026-08-12 (Estimated); Study Completion 2027-02-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | 1 month after the surgery
  Rate of pathologic complete response (pCR) after surgery

SECONDARY OUTCOMES:
Grade 3-4 adverse effects rate | From the date of randomization until 3 months after the completion neoadjuvant therapy
  Rate of chemotherapy, radiotherapy and immunotherapy related adverse events
Anal function | From the date of randomization until 36 months after the surgery
  Anal function will be evaluated using LARS score
Surgical complication | The surgical complications were assessed within 3 months after the surgery
  Rate of surgical complications, such as intraoperative hemorrhage, anastomotic leakage, intestinal obstruction, etc.
3-year local recurrence free survival (LRFS) rate | From the date of randomization until the date of first documented pelvic failure, assessed up to 36 months
  Rate of 3-year local recurrence free survival
3-year disease free survival (DFS) rate | From the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Rate of 3-year disease free survival
3-year overall survival (OS) rate | From the date of randomization until the date of death from any cause, assessed up to 36 months
  Rate of 3-year overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China